CLINICAL TRIAL: NCT05244512
Title: Online Training to Improve Evidence-based Leadership Competencies Among Nurse Leaders in Finland: Study Protocol for a Randomised Feasibility Trial (EVILED-FI)
Brief Title: Evidence-based Leadership in Nurse Leaders-FI
Acronym: EVILEAD-FI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turku (Other)
Collaborators: Central South University (Other); Sichuan University (Other); Swinburne University of Technology (Other)
Responsible Party: Principal Investigator, Maritta Välimäki, Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UTUEvidence
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Leadership
Keywords: feasibility, randomised controlled trial, training

STUDY DESIGN:
Intervention Model Description: A single-blind, individually randomised, two-arm parallel-group controlled feasibility trial design will be used.
Who Masked: Participant, Care Provider
Masking Description: Tutors and researchers involved in the screening and baseline assessment will not be blind to the interventions provided during the trial. Participants, care providers and statistician will be kept blind to the study conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-based leadership training (Experimental): The training course will take 6 months. It is divided into seven online modules. Participants join the course based on pre-structured schedule. The progress of the training course will follow specific steps to improve participants' evidence-based leadership competencies. First, each participant identifies one leadership problem on daily practice. Second, organisational data will be collected and analysed to increase the understanding of the key problem. Third, scientific literature will be searched, identified and critically appraised to find solutions. Fourth, the views of stakeholders (patients, clinicians, family members, etc.) are considered together with ethical implications. And last, all sources of information are critically appraised, new solution will be designed and implemented into the practice, and evaluated in real world context. Each module includes specific learning material. Trained tutors are responsible for mentoring each module.
  Interventions: Other: Evidence-based leadership training
- Conventional training (Active Comparator): The participants will join a training course with the same structure, topics, and timing as the experimental group. However, training in this group is based on independent learning methods. The participants have access to the separate learning platform, which includes reading material to be read independently. No group discussions with peers, self-reflection, assignments, or support from tutors will be offered.
  Interventions: Other: Conventional training

INTERVENTIONS:
Other: Evidence-based leadership training — 7-modules online training over six months mentored by tutors. Independent familiarisation of reading material, peer-group discussions, self-reflection, assignments, tutor's feedback.
  Arms: Evidence-based leadership training
Other: Conventional training — 7-modules online training over six months. Independent reading only.
  Arms: Conventional training

SUMMARY:
This study protocol describes a randomised feasibility trial that will evaluate the feasibility and preliminary effectiveness of the training course to improve evidence-based leadership competencies among nurse leaders working in hospitals in Finland.

DETAILED DESCRIPTION:
This study will include a 6-months training intervention for nurse leaders working in hospital settings in Finland. About 140 nurse leaders fulfilling the eligibility criteria will be randomly allocated (1:1) to participate in the online training course about evidence-based leadership or conventional leadership training course (reading material only).

ELIGIBILITY:
Inclusion Criteria:

* Official managerial role in the study organisation (hospital, clinic, ward level), which give them an authority to act as a nurse leader and monitor, develop and evaluate the care
* Being in full time or part time position
* All sex
* Aged up to 65 years
* Working in the study sites at the time of the recruitment
* Ability to read and write Finnish language
* Willingness to join the study based on their own free will
* Informed consent obtained

Exclusion Criteria:

* Non-nursing professionals in leadership position (e.g. physician, psychologist, pharmacist, dietician/nutritionist, dentist, physiotherapist, radiation therapist, paramedic, occupational therapist, social worker, or disability worker)
* Speaking only other languages than Finnish (e.g. Swedish or English)
* Out of duty during the recruitment period for family leave, long term sick leave, study leave or any other reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the intervention | 6 months
  The degree of execution (success and failure of execution) of the intervention protocol by calculating the number of logins for each module and all participants
Adherence in the course | 6 months
  Adherence in the course by calculating the number of returned course tasks out of all possible tasks
Adherence in the course tasks | 6 months
  Adherence in the course by calculating the number of returned course tasks by each participant
Drop-out rate | 6 months
  The drop-out rate calculated by the number of participants who left the study early (no follow-up data)

SECONDARY OUTCOMES:
Acceptability in recruitment | Baseline
  The number of nurse leaders who accepted (or refused) the invitation to participate in the research study
Feasibility of the eligibility criteria | Baseline
  The number of nurse leaders who fulfilled eligibility criteria
Feasibility of the outcome instruments for measuring the potential effectiveness of the online course | Baseline and 6 months
  The number of missing variables of each returned instrument
Leadership skills (Multifactor Leadership Questionnaire [MLQ]) | Baseline and 6 months
  Multifactor Leadership Questionnaire (MLQ)
Evidence-based practice, knowledge, and attitudes (Evidence Based Practice Questionnaire [EBPQ]) | Baseline and 6 months
  Evidence-Based Practice Questionnaire (EBPQ)
Self-efficacy (General Self-Efficacy Scale [GSE]) | Baseline and 6 months
  General Self-Efficacy Scale (GSE)
Self-esteem (Rosenberg Self-Esteem Scale [RSE]) | Baseline and 6 months
  Rosenberg Self-Esteem Scale (RSE)
Intention to leave (questionnaire) | Baseline and 6 months
  Three-item questionnaire
Course feedback | 6 months
  Eight-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maritta A Välimäki, Principal Investigator — University of Turku
Locations (1):
- Helsingin kaupunki, psykiatria, Helsinki, South Finland, Finland

IPD SHARING:
Plan to Share IPD: No
According to the ethical reasons

REFERENCES:
- [Derived] Valimaki MA, Kirsi H, Yang M, Lantta T, Varpula J, Liu G, Tang Y, Chen W, Hu S, Chen J, Loyttyniemi E, Li X. Online training to improve evidence-based leadership competencies among nurse leaders in Finland and China: study protocols for two randomised feasibility trials. BMJ Open. 2023 Aug 14;13(8):e067306. doi: 10.1136/bmjopen-2022-067306. PMID 37580090

DOCUMENTS (1):
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT05244512/ICF_000.pdf